CLINICAL TRIAL: NCT00981084
Title: The Impact of Armodafinil on Neurocognition and Cognitive Fatigue in Multiple Sclerosis: a Double-Blind Randomized Crossover Study
Brief Title: Impact of Armodafinil on Neurocognition and Cognitive Fatigue in Multiple Sclerosis (MS)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Missouri, Kansas City (Other)
Collaborators: University of Kansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: C10953/6113
Record Dates: First submitted 2009-09-18; First posted 2009-09-22 (Estimated); Results first posted 2013-10-14 (Estimated); Last update posted 2013-10-14 (Estimated); Status verified 2013-08

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- armodafinil and placebo (Experimental): All participants will receive one dose of armodafinil and one dose of placebo in a cross-over design
  Interventions: Drug: armodafinil

INTERVENTIONS:
Drug: armodafinil — Half of the patients will be randomized to receive a single oral dose of placebo prior to the first testing session. After a washout period of one week, they will then receive 250mg of armodafinil prior to a second testing session (P/A group). The other half of patients will be randomized to receive the active drug first. After a washout period of one week, they will receive the placebo prior to a second testing session (A/P group). As plasma levels of armodafinil peak between 2-4 hours after administration, participants will be asked to take a single 250mg capsule 2 hours prior to the scheduled testing sessions.
  Other Names: NuVigil

SUMMARY:
The investigation will involve a double-blind, placebo controlled, cross-over study examining the efficacy of armodafinil in improving neurocognitive functioning and reducing cognitive fatigue in MS. Patients who report MS-related cognitive difficulties and perform at least 1 standard deviation below the mean on a brief cognitive screen will be given a thorough neuropsychological evaluation at two time points. Half of the patients will be randomized to receive a single oral dose of lactose placebo prior to the first testing session. After a washout period of one week, they will then receive 250mg of armodafinil prior to a second testing session (P/A group). The other half of patients will be randomized to receive the active drug first. After a washout period of one week, they will receive the placebo prior to a second testing session (A/P group). As plasma levels of armodafinil peak between 2-4 hours after administration, participants will be asked to take a single 250mg capsule 2 hours prior to the scheduled testing sessions.

ELIGIBILITY:
Inclusion Criteria:

* relapsing remitting and secondary progressive MS patients
* between the ages of 18 and 60
* report cognitive difficulties.
* perform 1 sd or more below cut-off on cognitive screening measure

Exclusion Criteria:

* no history of alcohol/drug abuse or nervous system disorder other than MS
* no sensory impairments that might interfere significantly with cognitive testing
* no developmental history of learning disability or attention-deficit/hyperactivity disorder
* no medical condition other than MS that could substantially affect cognition
* no relapse and/or corticosteroid use within four weeks of assessment;
* no current use of modafinil, armodafinil or other psychostimulants.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2009-09; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jared M Bruce, PhD, Principal Investigator — University of Missouri, Kansas City; Sharon Lynch, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who demonstrated at least mild cognitive impairment on a screening measure were recruited from a large MS neurology clinic in the Midwest from 2009 to 2011.
Groups:
- Armodafinil First and Placebo Second: Patients randomly assigned to this condition received a 250 mg dose of armodafinil in the first treatment period. There was then a one week washout period. They received a placebo in the second treatment period. Testing was conducted 2 hours after treatment adminsitration using counterbalanced alternate forms.
- Placebo First and Armodafinil Second: Patients randomly assigned to this condition received a placebo in the first treatment period. There was then a one week washout period. They then received 250 mg armodafinil in the second treatment period. Testing was conducted 2 hours after treatment adminsitration using counterbalanced alternate forms.
Period: First Intervention (One Day)
Arm/Group | Armodafinil First and Placebo Second | Placebo First and Armodafinil Second
Started | 16 | 17
Completed | 16 | 17
Not Completed | 0 | 0
Period: Washout Period (7 Days)
Arm/Group | Armodafinil First and Placebo Second | Placebo First and Armodafinil Second
Started | 16 | 17
Completed | 16 | 17
Not Completed | 0 | 0
Period: Second Intervention (One Day)
Arm/Group | Armodafinil First and Placebo Second | Placebo First and Armodafinil Second
Started | 16 | 17
Completed | 16 | 17
Not Completed | 0 | 0
Period: Post Intervention (Data Analysis)
Arm/Group | Armodafinil First and Placebo Second | Placebo First and Armodafinil Second
Started | 16 | 17
Completed | 14 | 16
Not Completed | 2 | 1
Not completed — poor effort | 1 | 1
Not completed — imbalance in disease subtype | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Armodafinil Then Placebo: All participants will receive one dose of armodafinil and one dose of placebo in a cross-over design
  armodafinil : Half of the patients will be randomized to receive a single oral dose of placebo prior to the first testing session. After a washout period of one week, they will then receive 250mg of armodafinil prior to a second testing session (P/A group). The other half of patients will be randomized to receive the active drug first. After a washout period of one week, they will receive the placebo prior to a second testing session (A/P group). As plasma levels of armodafinil peak between 2-4 hours after administration, participants will be asked to take a single 250mg capsule 2 hours prior to the scheduled testing sessions.
- Total: Total of all reporting groups
Arm/Group | Armodafinil Then Placebo | Placebo Then Armodafinil | Total
Number analyzed (Participants) | 16 | 17 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 17 | 33
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 47.71 (5.89) | 49.94 (7.22) | 49.15 (6.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 15 | 28
  Male | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 16 | 17 | 33

OUTCOME MEASURES:

1. Primary Outcome: Learning and Memory Measures.
Description: Testing was completed after first intervention and again after second intervention.
  Higher scores indicate better performance. Scores from derived by subtracting session 2 scores from session 1 scores.
  Rey Auditory Verbal Learning Test (RAVLT)- Measure of Verbal Learning (Min = 0; Max = 75).
  RAVLT Delay - Measure of Delayed Verbal Recall (Min = 0; Max = 15).
  Brief Visuospatial Memory Test (BVMT) Learning - Measure of Visual Learning (Min = 0; Max = 36).
  BVMT Delay - Measure of Delayed Visual Recall (Min = 0; Max = 12).
Time Frame: Outcome was assessed after each intervention (2 time points). Time 2 scores were subtracted from time 1 scores.
Measure: Mean (Standard Deviation); unit: Items recalled
Groups:
- Placebo/Armofafinil: placebo first then armodafinil. Participants were tested after each intervention with alternate forms of outcome measures. Outcome scores from session 2 were subtracted from session 1 scores.
- Armodafinil/Placebo: armodafinil first and then placebo. Participants were tested after each intervention with alternate forms of outcome measures. Outcome scores from session 2 were subtracted from session 1 scores.
Arm/Group | Placebo/Armofafinil | Armodafinil/Placebo
Number analyzed (Participants) | 16 | 14
Items recalled
  Auditory Verbal Learning Test - Learning | -3.38 (7.32) | -.07 (6.06)
  Aditory Verbal Learning Test Delay | -1.38 (1.89) | 1.93 (2.70)
  Brief Visuospatial Memory Test Learning | .88 (4.63) | -1.57 (5.71)
  Brief Visuospatial Memory Test Delay | .56 (1.50) | -.57 (2.17)
Statistical Analysis 1: Comparison: Placebo/Armofafinil vs Armodafinil/Placebo; We used a crossover design to exame whether a single dose of armodafinil would improve cognition in MS. For hypothesis testing analyses, we used a statistical approach that accounts for period (session) effects. We subtracted session 2 performance from session 1 performance on the RVLT learning, yeilding a difference score. we conducted an independent samples t test with treatment order as the independent variable (A/P vs. P/A) and the difference score as the dependent variable; Test type: Superiority or Other; p = .19, t-test, 2 sided
Statistical Analysis 2: Comparison: Placebo/Armofafinil vs Armodafinil/Placebo; We used a crossover design to exame whether a single dose of armodafinil would improve cognition in MS. For hypothesis testing analyses, we used a statistical approach that accounts for period (session) effects. We subtracted session 2 performance from session 1 performance on the RVLT delay, yielding a difference score. we conducted an independent samples t test with treatment order as the independent variable (A/P vs. P/A) and the difference score as the dependent variable; Test type: Superiority or Other; p = .0005, t-test, 2 sided
Statistical Analysis 3: Comparison: Placebo/Armofafinil vs Armodafinil/Placebo; We used a crossover design to exame whether a single dose of armodafinil would improve cognition in MS. For hypothesis testing analyses, we used a statistical approach that accounts for period (session) effects. We subtracted session 2 performance from session 1 performance on the BVMT learning, yeilding a difference score. we conducted an independent samples t test with treatment order as the independent variable (A/P vs. P/A) and the difference score as the dependent variable; Test type: Superiority or Other; p = .21, t-test, 2 sided
Statistical Analysis 4: Comparison: Placebo/Armofafinil vs Armodafinil/Placebo; We used a crossover design to exame whether a single dose of armodafinil would improve cognition in MS. For hypothesis testing analyses, we used a statistical approach that accounts for period (session) effects. We subtracted session 2 performance from session 1 performance on the BVMT delay, yielding a difference score. we conducted an independent samples t test with treatment order as the independent variable (A/P vs. P/A) and the difference score as the dependent variable; Test type: Superiority or Other; p = .10, t-test, 2 sided

2. Primary Outcome: CPT -Test of Information Processing Speed
Description: Lower scores indicate better perforamnce. Scores from derived by subtracting session 2 scores from session 1 scores.
  Continuous Performance Test (CPT) - Vigilance and reaction time.
Time Frame: Outcome was assessed after each intervention (2 time points). Time 2 scores were subtracted from time 1 scores.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo/Armofafinil | Armodafinil/Placebo
Number analyzed (Participants) | 16 | 14
milliseconds | -1.18 (37.62) | 15.04 (50.30)
Statistical Analysis 1: Comparison: Placebo/Armofafinil vs Armodafinil/Placebo; We used a crossover design to exame whether a single dose of armodafinil would improve cognition in MS. For hypothesis testing analyses, we used a statistical approach that accounts for period (session) effects. We subtracted session 2 performance from session 1 performance on the CPT, yielding a difference score. we conducted an independent samples t test with treatment order as the independent variable (A/P vs. P/A) and the difference score as the dependent variable; Test type: Superiority or Other; p = .33, t-test, 2 sided

3. Primary Outcome: Stroop
Description: Stroop - Test of impulsivity (min = 0, max = none). Higher scores indicate better performance. Scores from derived by subtracting session 2 scores from session 1 scores.
Time Frame: Outcome was assessed after each intervention (2 time points). Time 2 scores were subtracted from time 1 scores.
Measure: Mean (Standard Deviation); unit: number of colors named
Arm/Group | Placebo/Armofafinil | Armodafinil/Placebo
Number analyzed (Participants) | 16 | 14
number of colors named | -1.69 (3.38) | -2.86 (3.72)
Statistical Analysis 1: Comparison: Placebo/Armofafinil vs Armodafinil/Placebo; We used a crossover design to examine whether a single dose of armodafinil would improve cognition in MS. For hypothesis testing analyses, we used a statistical approach that accounts for period (session) effects. We subtracted session 2 performance from session 1 performance on the Stroop, yielding a difference score. We conducted an independent samples t-test with treatment order as the independent variable (A/P vs. P/A) and the difference score as the dependent variable; Test type: Superiority or Other; p = .37, t-test, 2 sided

4. Primary Outcome: Word Generation
Description: Word Generation - Measure of verbal fluency. (Min = 0; No Max. )Higher scores indicate better performance. Scores from derived by subtracting session 2 scores from session 1 scores.
Time Frame: Outcome was assessed after each intervention (2 time points). Time 2 scores were subtracted from time 1 scores.
Measure: Mean (Standard Deviation); unit: number of words generated
Arm/Group | Placebo/Armofafinil | Armodafinil/Placebo
Number analyzed (Participants) | 16 | 14
number of words generated | -.69 (5.21) | -1.71 (3.24)
Statistical Analysis 1: Comparison: Placebo/Armofafinil vs Armodafinil/Placebo; We used a crossover design to examine whether a single dose of armodafinil would improve cognition in MS. For hypothesis testing analyses, we used a statistical approach that accounts for period (session) effects. We subtracted session 2 performance from session 1 performance on the Word Generation, yielding a difference score. We conducted an independent samples t-test with treatment order as the independent variable (A/P vs. P/A) and the difference score as the dependent variable; Test type: Superiority or Other; p = .53, t-test, 2 sided

ADVERSE EVENTS:
Groups:
- Placebo Then Armodafinil (Placebo): Adverse events reported after taking placebo in the Placebo then Armodafinil Group
- Armodafinil Then Placebo (Armodafinil): Adverse events reported after taking armodafinil in the Armodafinil then placebo group
- Placebo Then Armodafinil (Armodafinil): Adverse events following armodafinil in the placebo/armodafinil group
- Armodafinil Then Placebo (Placebo): number of adverse events following placebo in the armodafniil then placebo condition.
Arm/Group | Placebo Then Armodafinil (Placebo) | Armodafinil Then Placebo (Armodafinil) | Placebo Then Armodafinil (Armodafinil) | Armodafinil Then Placebo (Placebo)
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/16 | 0/17 | 0/16
Other Adverse Events (participants affected / at risk) | 2/17 | 3/16 | 2/17 | 1/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Then Armodafinil (Placebo) (N=17) | Armodafinil Then Placebo (Armodafinil) (N=16) | Placebo Then Armodafinil (Armodafinil) (N=17) | Armodafinil Then Placebo (Placebo) (N=16)
sleep difficulties (Nervous system disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0) — participants reported some difficulty falling asleep
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
A small pilot trial with only one dose of drug administered. Limitations include the very small sample and the use of a single-dose cross-over design.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less